CLINICAL TRIAL: NCT00316836
Title: The Association of Breast Density Changes, Plasma Hormone Changes, and Breast Cancer Recurrence: A Companion Study to NCIC CTG MA.27
Brief Title: Breast Density, Hormone Levels, and Anticancer Drug Levels in Women With Invasive Breast Cancer Who Are Receiving Exemestane or Anastrozole
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Other Study IDs: NCCTG-N0434; NCCTG-N0434; CAN-NCIC-MA27D; CDR0000462330 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patients complete a 10-minute questionnaire about factors that might affect changes in breast density at baseline and another questionnaire at 1 year and 2 years post registration. Blood samples are collected at baseline (before initiation of treatment ) and at 1 year post registration for hormone and drug level analysis. Mammograms taken prior to registration (within 12 months prior to enrollment) and at approximately 1 and 2 years post-registration to this study are retrieved and digitized for determination of percent breast density and dense area.
  Interventions: Procedure: mammography

INTERVENTIONS:
Procedure: mammography

SUMMARY:
RATIONALE: Understanding the relationship between breast density, levels of hormones in the blood, and levels of anticancer drugs in the blood may help improve the ability to plan effective treatment for women with invasive breast cancer.

PURPOSE: This clinical trial is studying the relationship between breast density and blood levels of hormones and anticancer drugs in women with invasive breast cancer who are receiving exemestane or anastrozole.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the change in percent breast density and dense area in response to aromatase inhibitor therapy from pretreatment to 1 year, 1 year to 2 years, and pretreatment to 2 years in women with invasive breast cancer.
* Determine the changes in percent breast density and dense area in response to aromatase inhibitor therapy from pretreatment to 1 year and correlate the changes with changes in plasma hormones (e.g., estrone, estrone-sulfate, estradiol, and sex hormone binding globulin) and drug levels (anastrozole or exemestane) over the same period in women with invasive breast cancer.
* Determine the change over time in percent breast density and dense area (from pretreatment to the time period prior to local recurrence) in the contralateral breast in correlation to local recurrence of breast cancer.

Secondary

* Determine the change over time in percent breast density and dense area in the contralateral breast in correlation to the development of contralateral breast cancer.
* Determine whether women with high pretreatment percent density (upper tertile) experience greater decreases in percent breast density at 1 and 2 years of aromatase inhibitor therapy than women with low pretreatment percent density (lower tertile).
* Determine whether women with high pretreatment dense area (upper tertile) experience greater decreases in dense area at 1 and 2 years of aromatase inhibitor therapy than women with low pretreatment dense area (lower tertile).
* Correlate haplotype tagged single nucleotide polymorphisms in genes in the aromatase pathway (identified thorough the Mayo Clinic and Indiana University Pharmacogenomics Research Network Projects) with changes in percent and area breast density, plasma hormone levels, and 1-year drug levels.

OUTLINE: This is a multicenter, companion study.

Patients complete a 10-minute questionnaire about factors that might affect changes in breast density at baseline and another questionnaire at 1 year and 2 years post registration. Blood samples are collected at baseline (before initiation of treatment ) and at 1 year post registration for hormone and drug level analysis. Mammograms taken prior to registration (within 12 months prior to enrollment) and at approximately 1 and 2 years post-registration to this study are retrieved and digitized for determination of percent breast density and dense area.

PROJECTED ACCRUAL: A total of 550 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer
* Completely resected disease
* One intact, noncancerous breast with no prior breast surgery in that breast except breast biopsy

  * Mammogram available taken within 12 months prior to enrollment that includes side- and top-down views of the intact, noncancerous breast
* Estrogen receptor- and/or progesterone receptor-positive tumor

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal
* Agrees to retrieve and digitize mammograms taken prior to registration (within 12 months prior to atudy entry) and at approximately 1 and 2 years post-registration to this study
* Agrees to have an additional blood banking specimen drawn at the same time as pre-treatment specimens are drawn for parent protocol CAN-NCIC-MA27
* Agrees to have blood sample taken at 12 months post-registration on this study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 6 months since prior hormone replacement therapy, oral contraceptives, tamoxifen, raloxifene, other selective estrogen-receptor modulators, or gonadotropin releasing-hormone analogues before pre-registration mammogram

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed with breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 554 (Actual)
Dates: Start 2006-04; Primary Completion 2010-10 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Changes in breast density measured by percent and area at 1 and 2 years | Up to 2 years
Correlation of changes in breast density with plasma hormones and drug levels measured by estrone, estrone-sulfate, estradiol, sex hormone binding globulin, anastrozole, or exemestane levels at 1 and 2 years | Up to 2 years

SECONDARY OUTCOMES:
Correlation of breast density with contralateral breast cancers at 1 and 2 years | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James N. Ingle, MD, Study Chair — Mayo Clinic
Locations (324):
- United States (311):
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Peninsula Medical Center, Burlingame, California
  - North Bay Cancer Center, Fairfield, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - California Cancer Care, Incorporated - Greenbrae, Greenbrae, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health - Western Division Cancer Research Group, Greenbrae, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - West Florida Cancer Institute at West Florida Hospital - Pensacola, Pensacola, Florida
  - Augusta Oncology Associates - Walton Way, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Kootenai Cancer Center - Coeur d'Alene, Coeur d'Alene, Idaho
  - Snake River Oncology of Eastern Idaho PLLC, Idaho Falls, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Delnor Community Hospital - Geneva, Geneva, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Bloomington Hospital Regional Cancer Institute, Bloomington, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Community Hospital, Munster, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Heartland Oncology and Hematology, Council Bluffs, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, PC - West Ridgeway Avenue, Waterloo, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Central Maine Comprehensive Cancer Center at Central Maine Medical Center, Lewiston, Maine
  - Mercy Hospital, Portland, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - NSMC Cancer Center - Peabody, Peabody, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Oncology Care Associates, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Fergus Falls, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - St. Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Warren Hospital, Phillipsburg, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Finger Lakes Hematology and Oncology, Clifton Springs, New York
  - Adirondack Cancer Care - Glens Falls, Glens Falls, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Cleo Craig Cancer Research Clinic, Lawton, Oklahoma
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Cancer Center at Phoenixville Hospital, Phoenixville, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - CCOP - Scott and White Hospital, Temple, Texas
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Valley Medical Center, Renton, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Central Wisconsin Cancer Program at Agnesian HealthCare, Fond du Lac, Wisconsin
  - Oncology Alliance, SC - Milwaukee - East, Glendale, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Medical Consultants, Limited, Milwaukee, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Canada (13):
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Cambridge Memorial Hospital, Cambridge, Ontario
  - Algoma District Cancer Program at Sault Area Hospital, Sault Ste. Marie, Ontario
  - Cancer Care Program at Thunder Bay Regional Health Sciences, Thunder Bay, Ontario
  - Edmond Odette Cancer Centre at Sunnybrook, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Hopital du Saint-Sacrement - Quebec, Québec, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan